CLINICAL TRIAL: NCT04172194
Title: Endoarterial Treatment in Combination With Percutaneous Thermoablation for Medium-sized and Oligonodular Hepatocellular Carcinomas
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-PT-02
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PT Group: patients with hepatocellular carcinoma treated by percutaneous thermoablation alone
- PT+TAC group: patients with hepatocellular carcinoma treated by pecutaneous thermoablation comined in a single session with trans-arterial chemoembolization

SUMMARY:
Background: The association of transcatheter arterial chemotherapy infusion (TAC) with percutaneous ablation (PT) has been introduced as a method to increase the ablative zone. The aim of this study was to evaluate the efficacy of PT and TAC performed in a single session for HCCs between 30 and 50 mm or oligonodular up to 30 mm.

Methods: Thirty patients with a histologically proven HCC, uninodular between 30 and 50 mm or oligonodular (n≤3) up to 30 mm, treatment-naïve and non-metastatic, received combination treatment ("PT+TAC group"). A "control" group consisted of 34 patients with uninodular HCC up to 30 mm without any poor prognostic criteria treated with PT alone ("PT group").

ELIGIBILITY:
Inclusion Criteria:

- hepatocellular carcinoma pouved by pathology,

Exclusion Criteria:

- metastases

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
overall survival | 30 minutes
  death

SECONDARY OUTCOMES:
relapse free survival | 30 minutes
  relapse
tolerance | 30 minutes
  apparition of complication define by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No